CLINICAL TRIAL: NCT03733158
Title: Comparison of the New Flexible Tip Bougie Catheter and Standard Bougie Stylet for Tracheal Intubation by Anesthesiologists in Different Difficult Airway Scenarios: a Randomized Crossover Trial
Brief Title: Flexible Tip Bougie Catheter Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lazarski University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: INT_2018_UL
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Emergency Medicine; Endotracheal Intubation; Cardiopulmonary Arrest
Keywords: endotracheal intubation; emergency medicine; cardiopulmonary resuscitation; physician
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Normal airway (Experimental): intubation in normal aurway condition
  Interventions: Device: the standard Bougie stylet for difficult intubation; Device: The new Flexible Tip Bougie catheter
- Tongue edema (Experimental): intubation in Tongue edema condition
  Interventions: Device: the standard Bougie stylet for difficult intubation; Device: The new Flexible Tip Bougie catheter
- Pharyngeal obstruction (Experimental): intubation in Tongue edema condition
  Interventions: Device: the standard Bougie stylet for difficult intubation; Device: The new Flexible Tip Bougie catheter
- Manual cervical inline stabilization (Experimental): intubation in Manual cervical inline stabilization condition
  Interventions: Device: the standard Bougie stylet for difficult intubation; Device: The new Flexible Tip Bougie catheter
- Cervical collar stabilization (Experimental): intubation in Cervical collar stabilization condition
  Interventions: Device: the standard Bougie stylet for difficult intubation; Device: The new Flexible Tip Bougie catheter
- Cervical collar stabilization and pharyngeal obstruction (Experimental): intubation in Cervical collar stabilization and pharyngeal obstruction condition
  Interventions: Device: the standard Bougie stylet for difficult intubation; Device: The new Flexible Tip Bougie catheter

INTERVENTIONS:
Device: the standard Bougie stylet for difficult intubation — intubation with the standard Bougie stylet for difficult intubation and endotracheal tube 7.0 internal diameter
Device: The new Flexible Tip Bougie catheter — intubation with The new Flexible Tip Bougie catheter and endotracheal tube 7.0 internal diameter

SUMMARY:
We, therefore conducted a randomized cross over study to evaluate the usefulness of this new device use by experienced anesthesiologists in several airway manikin scenarios. We hypothesized that in the hands of experienced anesthesiologists the new Flexible Tip Bougie catheter would perform comparably to the standard bougie catheter) in the normal airway scenario. In the difficult airway (both tongue edema, manual in-line stabilization, or cervical collar stabilization), we hypothesized that the new Flexible Tip Bougie catheter would prove superior to the standard Bougie stylet.

ELIGIBILITY:
Inclusion Criteria:

* physicians
* give voluntary consent to participate in the study
* none experience in videolaryngoscopy
* less than 1 year experience in medicine

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
time to intubation | 1 day
  time from pick up device to the final placement tube in trachea

SECONDARY OUTCOMES:
success of intubation | 1 day
  A failed intubation attempt was defined as an attempt in which the trachea was not intubated, or which required more than 120 seconds to perform
Number of optimalization maneuvers | 1 day
  the number of optimization maneuvers required (re-adjustment of head position, second assistant) to aid endotracheal intubation.
Ease of use | 1 day
  self-reported percentage the vocal cord visualization. A 100% score is a extremely difficult procedure. A Ease of use score of 1% means that procedure is extremely easy
Dental compression | 1 day
  An independent observer scored the severity of dental compressions, which was calculated based on the number of audible teeth clicks (0; 1; ≥2) with the Laerdal airway trainer, and based on a grading of pressure of the teeth (none = 0; mild = 1; moderate/serve ≥2) on the Simman®3G simulator. At the end of each scenario, each participant scored the ease of use of each intubation method on a visual analogue scale (VAS; from 0=Extremely Easy to 100=Extremely Difficult).

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Phd, Principal Investigator — Lazarski University
Locations (1):
- Lazarski University, Warsaw, Masovia, Poland

IPD SHARING:
Plan to Share IPD: Undecided
data will be available from the main investigator

REFERENCES:
- [Derived] Ruetzler K, Smereka J, Abelairas-Gomez C, Frass M, Dabrowski M, Bialka S, Misiolek H, Plusa T, Robak O, Aniolek O, Ladny JR, Gorczyca D, Ahuja S, Szarpak L. Comparison of the new flexible tip bougie catheter and standard bougie stylet for tracheal intubation by anesthesiologists in different difficult airway scenarios: a randomized crossover trial. BMC Anesthesiol. 2020 Apr 20;20(1):90. doi: 10.1186/s12871-020-01009-7. PMID 32312225